CLINICAL TRIAL: NCT00206505
Title: A PHASE II STUDY OF THE CLINICAL AND BIOLOGIC EFFECTS OF DOCETAXEL (TAXOTERE) IN PATIENTS WITH LOCALLY ADVANCED BREAST CANCER
Brief Title: Neoadjuvant Taxotere
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Breast Care Center (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H 8448
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Neoadjuvant; Taxotere
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Taxotere

SUMMARY:
The purposes of this study are to better understand how Taxotere causes tumors to become smaller and to find out how effective Taxotere is in treating the type of breast cancer that you have.

DETAILED DESCRIPTION:
Systemic chemotherapy for operable breast cancer significantly decreases the risk of relapse and death. However, it is not possible to identify those patients at the outset who are likely to respond to adjuvant treatment and which type of treatment should be used. Adjuvant treatment given before surgery (neoadjuvant therapy) has a number of theoretical advantages in breast cancer, including a reduction in the requirement for mastectomy. Access to the primary tumor during early treatment allows for in vivo testing for change in molecular markers by repeat biopsies that may occur with successful treatment. Established prognostic factors like tumor size and nodal involvement are important indicators for breast cancer relapse and survival but have not been shown to be predictive of sensitivity to treatment. Estrogen receptor (ER) and progesterone receptor (PgR) expression predict for response to tamoxifen and endocrine treatment. However, predictive markers for chemotherapy are not established. Overexpression of c-erbB-2 has been associated with decreased response to CMF chemotherapy (cyclophosphamide, methotrexate, and 5-fluorouracil) in most studies. Accumulation of aberrant protein expressed by the mutated tumor suppressor gene p53 product may be associated with relative resistance to cytotoxic therapy. Tissue growth kinetics are determined by the balance between programmed cell death (apoptosis) and cell proliferation, and any alteration between the two may be regarded as a key element for the uncontrolled growth of malignant tumors. In vitro experiments suggest that many anti-cancer agents achieve their effect by inducing apoptosis. Mechanisms that suppress this process may, therefore, be important in the development of intrinsic and acquired chemotherapy resistance. A clinical study has reported an increase in labeled apoptotic leukemic cells during treatment. In breast cancer biopsy specimens, chemotherapy was found to induce apoptosis within the first 24 hours of treatment.

Measurement of biological molecular markers before and after exposure may, therefore, allow for early prediction of the likelihood of response to systemic therapy. Preoperative chemotherapy has been shown to result in changes in biomarkers, and these changes, when correlated with tumor response, may be early predictors of clinical outcome.

New treatment strategies are needed to improve the clinical outcome in breast cancer patients at high risk of recurrence. Even with the best present combination chemotherapy, radiotherapy, and surgery, disease recurrence and death is at least 60% in this population. Thus, new strategies are needed to improve survival. Recent advances that may improve clinical outcome include the use of taxoids (paclitaxel and docetaxel), a new class of cytotoxic agents, with reported higher response rates than standard anthracycline-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients must be female. 2. Signed informed consent. 3. Locally advanced breast cancers or primary breast cancers with concomitant metastatic disease are eligible. Locally advanced cancers must be of clinical and/or radiologic size >4 cm and/or are deemed surgically inoperable. 4. Negative serum pregnancy test within 7 days of starting study, if of child-bearing potential. 5. Adequate bone marrow function: Hematocrit of greater than 30%, total neutrophil count must be >1.5 x 10(9)/L and platelets of >100 x 10(9)/L prior to the start of any cycle. 6. Kidney function tests - within 1.5 times of the institution's upper limit of normal. Total serum bilirubin within upper limit of normal. 7. Electrocardiogram showing no acute ischemic changes. 8. Performance status (WHO scale) <2 (Appendix I) and life expectancy >1 year. 9. Age > 18 years. 10. No brain and/or leptomeningeal disease. 11. No previous or current malignancies at other sites within the last 5 years, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.

Exclusion Criteria:

* 1. Pregnancy or unwillingness to use reliable contraceptive method in women of child-bearing potential. 2. Severe underlying chronic illness or disease. 3. Peripheral neuropathy - grade 2 or greater. 4. Patients on other investigational drugs while on study will be excluded. 5. Severe or uncontrolled hypertension, history of congestive heart failure, or severe coronary arterial disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1999-01; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
efficacy of neoadjuvantTaxotere in patients with locally advanced breast cancer. Histological complete response rate

SECONDARY OUTCOMES:
biologic effects of docetaxel (Taxotere) by sequential core biopsies taken before and after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Chang, MD, Principal Investigator — Baylor Breast Center
Locations (1):
- Baylor Breast Center, Houston, Texas, United States

REFERENCES:
- See also: Web Site — http://www.breastcenter.tmc.edu